CLINICAL TRIAL: NCT00346710
Title: Communication Skills in Rheumatology Fellows
Brief Title: Patient Experiences in Rheumatology
Status: Withdrawn | Type: Observational
Why Stopped: Information was entered by mistake by a Research Assistant. Study never went beyond the initial discussion phase.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: NA_00001397
Record Dates: First submitted 2006-06-28; First posted 2006-06-30 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Rheumatic Disease
Keywords: communication; patient experience; fellowship training
MeSH Terms: conditions — Rheumatic Diseases; Communication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Information was entered by mistake by a Research Assistant. Study never went beyond the initial discussion phase.

ELIGIBILITY:
All adult patients who have an appointment scheduled at the Rheumatology Clinic at Good Samaritan Hospital, can speak and read English and are willing and capable of providing informed consent are eligible to participate. All fellows in the Rheumatology Fellowship training program will participate.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-06-01 (Actual); Primary Completion 2006-06-02 (Actual); Study Completion 2006-06-02 (Actual)

PRIMARY OUTCOMES:
Changes in patient and provider satisfaction scores will be measured at baseline and 6 months using self-report. | Baseline and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Clifton O Bingham, MD, Principal Investigator — Johns Hopkins University